CLINICAL TRIAL: NCT06604169
Title: An Observational Study of Subcutaneous Implantable Cardioverter Defibrillator in Patients with Hypertrophic Cardiomyopathy At High Risk of Sudden Cardiac Death
Status: Active, not recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: S-ICD in HCM
Record Dates: First submitted 2024-09-18; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HCM - Hypertrophic Cardiomyopathy; S-ICD System (implantable Defibrillator)
Keywords: HCM; S-ICD
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1. To observe the failure rate of S-ICD screening in HCM patients at high risk of SCD.
2. To observe the incidence of IAS in HCM patients with S-ICD implantation and explore the related factors of IAS.

DETAILED DESCRIPTION:
The study was a multicenter, prospective, observational study that prospectively included HCM patients assessed as meeting the ICD implantation indication at Fuwai Hospital and National Collaborative Hospitals from July 1, 2024 to June 30, 2027, for pre-operation screening of S-ICD, and follow-up of patients eventually implanted with S-ICD.

ELIGIBILITY:
Inclusion Criteria:

* HCM patients assessed as meeting the ICD implantation indication

Exclusion Criteria:

* Combined with bradycardia with pacing indications;
* Frequent monomorphic ventricular tachycardia require ATP therapy;
* With indications of CRT;
* Combined with other diseases, life expectancy is less than 1 year.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was a multicenter, prospective, observational study that prospectively included HCM patients assessed as meeting the ICD implantation indication at Fuwai Hospital and National Collaborative Hospitals from July 1, 2024 to June 30, 2027.
Sampling Method: Non-Probability Sample
Enrollment: 589 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
the failure rate of S-ICD screening | 3 months
  S-ICD screening failed
The inappropriate shock event | 3 months
  The incidence of inappropriate shock event

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: Undecided